CLINICAL TRIAL: NCT02619084
Title: Subthalamic Nucleus Deep Brain Stimulation in Tourette's Syndrome
Brief Title: Subthalamic Stimulation in Tourette's Syndrome
Acronym: STN-DBSinTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Luigi M. Romito, MD, PhD, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RF-131; GR-2009-1594645 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2015-10-02; First posted 2015-12-02 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Tourette's Syndrome; Tourette Syndrome; Gilles de la Tourette Syndrome; Tourette Disorder
Keywords: Tourette Syndrome; Subthalamic Nucleus; STN; Deep Brain Stimulation; DBS; Tic; Obsessive-compulsive disorders
MeSH Terms: conditions — Tourette Syndrome; Tics; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- STN DBS ON First (Experimental): The study will be performed according a randomized, double-blind, crossover design with two 3-month phases, during which the stimulation could be switched "on" or "off", separated by a 1-month washout period, At the end of the second double-blind phase, a further open period of 6 months with stimulation switched "on" will follow.
  Interventions: Procedure: STN DBS
- STN DBS OFF First (Experimental): The study will be performed according a randomized, double-blind, crossover design with two 3-month phases, during which the stimulation could be switched "on" or "off", separated by a 1-month washout period, At the end of the second double-blind phase, a further open period of 6 months with stimulation switched "on" will follow.
  Interventions: Procedure: STN DBS

INTERVENTIONS:
Procedure: STN DBS — Bilateral STN DBS
  Other Names: Deep Brain Stimulation of the subthalamic nucleus; Neurostimulators: Medtronic Activa® SC 37603; Extensions: Medtronic Model 37086; Leads: Medtronic Model 3389

SUMMARY:
The main objective of this project is to evaluate the efficacy of subthalamic nucleus deep brain stimulation (STN DBS) in treating motor and phonic tics in medically refractory Tourette's syndrome (TS).

Secondary objectives are to individuate and standardize the best electrical parameters for STN stimulation in TS, to evaluate the efficacy and safety on non-motor TS features, such as behavioral abnormalities and psychiatric disorders, during chronic STN stimulation, to correlate the improvement of TS motor and non-motor symptoms to the modification in brain activity recorded by PET study and to explore the pathophysiology of TS, and to evaluate the safety of STN DBS in TS patients.

DETAILED DESCRIPTION:
Background Tourette's syndrome (TS) is characterized by the occurrence, before 18 years of age, of multiple motor and vocal tics, which do not necessarily occur concomitantly. Tics constitute the clinical hallmark of TS; they are sudden, brief, intermittent involuntary (or semi-involuntary) movements (motor tics) or noises (sound tics). Tic severity is variable: some patients have mild or bearable tics, whereas in others tics are so severe to cause bone fractures or cervical myelopathy. Diagnostic criteria set by the Tourette Syndrome Classification Study Group and the American Psychiatric Association are commonly used. It is currently recognized that TS is far more common than previously thought, with a prevalence of 1 to 10 children of adolescents per 1000.

Tics are usually treated in cases where disability at school, in the social environment or at home is severe enough to warrant medical intervention. TS commonly presents with co-morbid features, mainly consisting in obsessive-compulsive traits, attention deficit with hyperactivity disorder and depression. Psychopathologic features are partly an aftermath of tics, particularly in those patients who display severe tics affecting their social and work activities. Therefore, amelioration of tics may substantially improve daily life and adaptation to social and work environments.

Medication is the first choice treatment, with the aim to reduce the intensity of tics and the associated clinical features. Different drugs, belonging to several pharmacologic classes, such as α-adrenergic drugs, typical and atypical neuroleptics, and tetrabenazine are used. In some cases drug treatment provides satisfactory symptomatic benefit. Overall, it is reckoned that a meaningful proportion of TS patients do not have adequate benefit with drug treatment and the majority of patients have side effects of variable severity.

Ablative psychosurgery has been historically used to treat more severe cases of TS, but the results have been disappointing and burdened by irreversible side effects. The recently developed technique of deep brain stimulation (DBS) allows to selectively modulate the activity of brain structures that control movements and behaviors in patients with different neurological disorders. This approach is warranted in those patients who respond poorly to available medical therapy.

Recently, therapeutic DBS trials have been performed in patients with severe TS, who were not satisfactorily controlled by medication. At first, the same thalamic nuclei targeted by ablative surgery, particularly the centromedian-parafascicular (CM-pf) nuclear complex, have been implanted with some success.

Another anatomical target has been the anterior capsule in proximity of the nucleus accumbens or the nucleus accumbens itself, aiming at interfering with tics and obsessive-compulsive features at the same time. More recently, the globus pallidus internum (GPi) has been implanted. This constitutes the main output station of the basal ganglia towards the thalamus and the cerebral cortex.

Hypothesis driven rationales

1. There is preliminary evidence that the subthalamic nucleus can be another promising target in treating motor and non-motor feature of TS. A clinical observation has recently shown that STN DBS improved motor and vocal tics in a patient with consistence of Parkinson's disease and TS
2. Literature evidences have showed that stereotyped behaviors in nonhuman primates, resembling tics and compulsive disorders, were related to dysfunction of the limbic parts of the globus pallidus externum, the STN, and the SN reticulata, rather than to dysfunction of the GPi
3. From a physiologic perspective, STN occupies a privileged position influencing both output nuclei of the basal ganglia, GPi and substantia nigra (SN) reticulata. Several findings have highlighted the putative role of the STN in integrating emotional, cognitive and motor functions and this nucleus would thus be an effective target for the treatment of conditions that combine motor symptoms, behavioral disorders, obsessive-compulsive disorders
4. Involvement of the SN in TS was also found in a functional MRI study. Furthermore, stimulation of the anterior STN was effective in reducing stereotypes in a primate model of behavioral disorder and STN DBS in PD can also result in behavioral changes. Indeed, the small size of this nucleus may allow modulation of abnormal neuronal activity of both limbic and sensorimotor territories, more easily than GPi or thalamic DBS
5. The small and well-defined volume of the STN combined with well standardized implant techniques, would lead to a reduced inter-patient variability in targeting

The novelty of the project The STN may be a potential target for DBS in TS. The choice of STN as a target for this project is the current model of basal ganglia functioning: this anatomical location aims at modulating the sensory-motor, associative and limbic subdivisions of cortico-subcortical-cortical loops that are thought to be dysfunctional in TS. STN DBS may provide a quicker relief of symptoms than medial thalamic nuclei or GPi stimulation.

The main objective of this project is to evaluate the efficacy of subthalamic nucleus deep brain stimulation (STN DBS) in treating motor and phonic tics in medically refractory Tourette's syndrome (TS).

Secondary objectives are to individuate and standardize the best electrical parameters for STN stimulation in TS, to evaluate the efficacy and safety on non-motor TS features, such as behavioral abnormalities and psychiatric disorders, during chronic STN stimulation, to correlate the improvement of TS motor and non-motor symptoms to the modification in brain activity recorded by PET study and to explore the pathophysiology of TS, and to evaluate the safety of STN DBS in TS patients.

Clinical evaluation will include a complete neurological examination (videotaped tic scales throughout), a structured psychological interview and a psychiatric evaluation. Quantitative evaluations will be performed using appropriate validated neurological (including the Yale Tic Global Severity Scale (YTGSS) and neuropsychological rating scales, including the Yale-Brown Obsessive Compulsive scale (Y-BOCS), as detailed hereafter.

Neurological evaluations

* Tourette's motor and phonic tics checklist
* YTGSS
* Global assessment scale (GAS)
* Global Clinical Impression Scale (GCI-S)
* Sickness Impact Profile (SIP)
* Gilles de la Tourette syndrome-quality of life scale (GTS-QOL)

Behavioral evaluations

* Y-BOCS
* Depression (MADRS, HAM-D)
* ADHD and Anxiety (ADHD-RS, HAM-A)

Neuropsychological evaluations

* Global deterioration
* Executive functions
* Working memory
* Fluency

Power calculation. A retrospective analysis of published data on DBS-treated TS patients reports an average YGTSS at inclusion of 50 ±15 points. This is in keeping with our inclusion criteria of YGTSS >35. Considering a 50% improvement as meaningful, a 25-point variation is expected from baseline to post-implant in the active stimulation group and a 10% 5-point variation in the sham stimulation group. The investigators assume a comparable standard deviation at baseline and at end of the observational periods and a good correlation of YGTSS measures (correlation coefficient: 0.8). An actual number of at least 5 patients per group should allow to demonstrate a 25-point YGTSS difference between the two active stimulation and the sham stimulation groups, with a statistical potency of 85% (bilateral Mann-Whitney-Wilcoxon test, alpha = 5 %).

ELIGIBILITY:
Inclusion Criteria:

* Age at least of 18 years (with potential exceptions)
* Diagnosis of TS based on the diagnostic criteria of the Tourette Syndrome Classification Study Group
* A Yale Tic Global Severity Scale (YTGSS) > 35/50 for at least 12 months, with tic severity documented by a standardized videotape assessment
* Inadequate response to standard drug treatment or botulinum toxin

Exclusion Criteria:

* Diagnosis of secondary tic disorder, of heredodegenerative or neurometabolic diseases or history of toxic exposures or encephalitis
* Previous surgery for TS (with potential exceptions)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Yale Global Tic Severity Scale | Three months after stimulation switched ON v pre-operative condition
  Primary outcome measure will evaluate the efficacy of subthalamic nucleus deep brain stimulation (STN DBS) in controlling motor and phonic tics (by evaluating the reduction on the Yale Global Tic Severity Scale - YGTSS) in patients with medically refractory Tourette syndrome (TS), in a study to be performed according a randomized, double-blind, crossover design with two 3-month phases, during which the stimulation could be switched "on" or "off", separated by a 1-month washout period.
  The assumption tested is that of a meaningful tic improvement by bilateral STN DBS (considered as ≥ 50% reduction in Yale Global Tic Severity Scale - YGTSS from baseline to post-implant in the active stimulation group). YGTSS is a semistructured clinician-rated instrument that assesses the severity and frequency of motor and phonic tics.

SECONDARY OUTCOMES:
Change in Milan Overall Dementia Assessment (MODA) | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects on TS neuropsychological features of STN stimulation. Assessments will be performed by administering the MODA (assessing specific neuropsychological tests, exploring the global deterioration, the executive functions, the working memory and fluency).
Change in brain activity recorded by PET | Three months after stimulation switched ON v pre-operative condition
  To correlate the improvement of TS motor and non-motor symptoms to the modification in brain activity recorded by PET study and to explore the pathophysiology of TS
STN DBS safety in treating medically-refractory Tourette syndrome | 24 months
  An analysis of adverse and side effects of surgery and STN stimulation will be performed during the whole observation period (24 months)
Change in Yale-Brown Obsessive Compulsive scale (Y-BOCS) | Three months after stimulation switched ON v pre-operative condition
  One of the secondary outcome will measure the effect of STN DBS in controlling obsessive-compulsive features (by evaluating the change on the Y-BOCS) in patients with medically refractory TS
Change in Global assessment scale (GAS). | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects of STN stimulation on the overall functioning of a TS subjects during the specified time period on a continuum from psychological or psychiatric sickness to health. Assessments will be performed by administering the GAS.
Change in Global Clinical Impression Scale (GCI-S) | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects of STN stimulation on the overall status of a TS subjects during the specified time period. Assessments will be performed by administering the GCI-S.
Change in Gilles de la Tourette syndrome-quality of life scale (GTS-QOL) | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects of STN stimulation on the overall QoL of a TS subjects during the specified time period. Assessments will be performed by administering the GTS-QOL.
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects of STN stimulation on the depressive features of a TS subjects during the specified time period. Assessments will be performed by administering the MADRS.
Change in ADHD Rating Scale-IV (ADHD-RS) | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects of STN stimulation on the ADHD symptoms of a TS subjects during the specified time period. Assessments will be performed by administering the ADHD-RS.
Change in Hamilton Anxiety Rating Scale (HAM-A) | Three months after stimulation switched ON v pre-operative condition
  To evaluate the effects of STN stimulation on the anxiety symptoms of a TS subjects during the specified time period. Assessments will be performed by administering the HAM-A.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi M Romito, MD, PhD, Principal Investigator — IRCCS Istituto Neurologico Carlo Besta, Milano, Italy
Locations (1):
- Fondazione IRCCS Istituto neurologico Carlo Besta, Milan, Milan, Italy

REFERENCES:
- [Background] de la Tourette G. Étude sur une affection nerveuse caractérisée par l'incoordination motrice accompagnée d'écholalie et de coprolalie. Arch Neurol 1885;9:158-200
- [Background] Jankovic J. Tourette's syndrome. N Engl J Med. 2001 Oct 18;345(16):1184-92. doi: 10.1056/NEJMra010032. No abstract available. PMID 11642235
- [Background] Leckman JF. Phenomenology of tics and natural history of tic disorders. Brain Dev. 2003 Dec;25 Suppl 1:S24-8. doi: 10.1016/s0387-7604(03)90004-0. PMID 14980368
- [Background] Fahn S. The clinical spectrum of motor tics. Adv Neurol. 1982;35:341-4. No abstract available. PMID 7148580
- [Background] Brill CB, Hartz WH, Mancall EL. Cervical disc herniation in the Gilles de la Tourette syndrome. Ann Neurol. 1981 Mar;9(3):311. doi: 10.1002/ana.410090323. No abstract available. PMID 6939410
- [Background] Definitions and classification of tic disorders. The Tourette Syndrome Classification Study Group. Arch Neurol. 1993 Oct;50(10):1013-6. doi: 10.1001/archneur.1993.00540100012008. PMID 8215958
- [Background] American Psychiatric Association. DSM-IV-TR Diagnostic and Statistical Manual of Mental Disorders, IV ed. Washington DC and London: 2000
- [Background] Kurlan R, McDermott MP, Deeley C, Como PG, Brower C, Eapen S, Andresen EM, Miller B. Prevalence of tics in schoolchildren and association with placement in special education. Neurology. 2001 Oct 23;57(8):1383-8. doi: 10.1212/wnl.57.8.1383. PMID 11673576
- [Background] Robertson MM. The prevalence and epidemiology of Gilles de la Tourette syndrome. Part 1: the epidemiological and prevalence studies. J Psychosom Res. 2008 Nov;65(5):461-72. doi: 10.1016/j.jpsychores.2008.03.006. Epub 2008 Oct 2. PMID 18940377
- [Background] Lombroso PJ, Scahill L. Tourette syndrome and obsessive-compulsive disorder. Brain Dev. 2008 Apr;30(4):231-7. doi: 10.1016/j.braindev.2007.09.001. Epub 2007 Oct 15. PMID 17937978
- [Background] Singer HS. Tourette's syndrome: from behaviour to biology. Lancet Neurol. 2005 Mar;4(3):149-59. doi: 10.1016/S1474-4422(05)01012-4. PMID 15721825
- [Background] Scahill L, Erenberg G, Berlin CM Jr, Budman C, Coffey BJ, Jankovic J, Kiessling L, King RA, Kurlan R, Lang A, Mink J, Murphy T, Zinner S, Walkup J; Tourette Syndrome Association Medical Advisory Board: Practice Committee. Contemporary assessment and pharmacotherapy of Tourette syndrome. NeuroRx. 2006 Apr;3(2):192-206. doi: 10.1016/j.nurx.2006.01.009. PMID 16554257
- [Background] Kenney C, Jankovic J. Tetrabenazine in the treatment of hyperkinetic movement disorders. Expert Rev Neurother. 2006 Jan;6(1):7-17. doi: 10.1586/14737175.6.1.7. PMID 16466307
- [Background] Silay YS, Jankovic J. Emerging drugs in Tourette syndrome. Expert Opin Emerg Drugs. 2005 May;10(2):365-80. doi: 10.1517/14728214.10.2.365. PMID 15934872
- [Background] de Divitiis E, D'Errico A, Cerillo A. Stereotactic surgery in Gilles de la Tourette syndrome. Acta Neurochir (Wien). 1977;(Suppl 24):73. doi: 10.1007/978-3-7091-8482-0_12. No abstract available. PMID 335809
- [Background] Rickards H, Wood C, Cavanna AE. Hassler and Dieckmann's seminal paper on stereotactic thalamotomy for Gilles de la Tourette syndrome: translation and critical reappraisal. Mov Disord. 2008 Oct 30;23(14):1966-72. doi: 10.1002/mds.22238. PMID 18792123
- [Background] Robertson M, Doran M, Trimble M, Lees AJ. The treatment of Gilles de la Tourette syndrome by limbic leucotomy. J Neurol Neurosurg Psychiatry. 1990 Aug;53(8):691-4. doi: 10.1136/jnnp.53.8.691. PMID 2213047
- [Background] Hassler R, Dieckmann G. [Stereotaxic treatment of tics and inarticulate cries or coprolalia considered as motor obsessional phenomena in Gilles de la Tourette's disease]. Rev Neurol (Paris). 1970 Aug;123(2):89-100. No abstract available. French. PMID 4932913
- [Background] Benabid AL, Chabardes S, Torres N, Piallat B, Krack P, Fraix V, Pollak P. Functional neurosurgery for movement disorders: a historical perspective. Prog Brain Res. 2009;175:379-91. doi: 10.1016/S0079-6123(09)17525-8. PMID 19660668
- [Background] Hardesty DE, Sackeim HA. Deep brain stimulation in movement and psychiatric disorders. Biol Psychiatry. 2007 Apr 1;61(7):831-5. doi: 10.1016/j.biopsych.2006.08.028. Epub 2006 Nov 27. PMID 17126303
- [Background] Mink JW, Walkup J, Frey KA, Como P, Cath D, Delong MR, Erenberg G, Jankovic J, Juncos J, Leckman JF, Swerdlow N, Visser-Vandewalle V, Vitek JL; Tourette Syndrome Association, Inc. Patient selection and assessment recommendations for deep brain stimulation in Tourette syndrome. Mov Disord. 2006 Nov;21(11):1831-8. doi: 10.1002/mds.21039. PMID 16991144
- [Background] Visser-Vandewalle V. DBS in tourette syndrome: rationale, current status and future prospects. Acta Neurochir Suppl. 2007;97(Pt 2):215-22. doi: 10.1007/978-3-211-33081-4_24. PMID 17691307
- [Background] Ackermans L, Temel Y, Visser-Vandewalle V. Deep brain stimulation in Tourette's Syndrome. Neurotherapeutics. 2008 Apr;5(2):339-44. doi: 10.1016/j.nurt.2008.01.009. PMID 18394575
- [Background] Vandewalle V, van der Linden C, Groenewegen HJ, Caemaert J. Stereotactic treatment of Gilles de la Tourette syndrome by high frequency stimulation of thalamus. Lancet. 1999 Feb 27;353(9154):724. doi: 10.1016/s0140-6736(98)05964-9. No abstract available. PMID 10073521
- [Background] Visser-Vandewalle V, Temel Y, Boon P, Vreeling F, Colle H, Hoogland G, Groenewegen HJ, van der Linden C. Chronic bilateral thalamic stimulation: a new therapeutic approach in intractable Tourette syndrome. Report of three cases. J Neurosurg. 2003 Dec;99(6):1094-100. doi: 10.3171/jns.2003.99.6.1094. PMID 14705742
- [Background] Servello D, Porta M, Sassi M, Brambilla A, Robertson MM. Deep brain stimulation in 18 patients with severe Gilles de la Tourette syndrome refractory to treatment: the surgery and stimulation. J Neurol Neurosurg Psychiatry. 2008 Feb;79(2):136-42. doi: 10.1136/jnnp.2006.104067. Epub 2007 Sep 10. PMID 17846115
- [Background] Houeto JL, Karachi C, Mallet L, Pillon B, Yelnik J, Mesnage V, Welter ML, Navarro S, Pelissolo A, Damier P, Pidoux B, Dormont D, Cornu P, Agid Y. Tourette's syndrome and deep brain stimulation. J Neurol Neurosurg Psychiatry. 2005 Jul;76(7):992-5. doi: 10.1136/jnnp.2004.043273. PMID 15965209
- [Background] Flaherty AW, Williams ZM, Amirnovin R, Kasper E, Rauch SL, Cosgrove GR, Eskandar EN. Deep brain stimulation of the anterior internal capsule for the treatment of Tourette syndrome: technical case report. Neurosurgery. 2005 Oct;57(4 Suppl):E403; discussion E403. doi: 10.1227/01.neu.0000176854.24694.95. PMID 16234657
- [Background] Burdick A, Foote KD, Goodman W, Ward HE, Ricciuti N, Murphy T, Haq I, Okun MS. Lack of benefit of accumbens/capsular deep brain stimulation in a patient with both tics and obsessive-compulsive disorder. Neurocase. 2010 Aug;16(4):321-30. doi: 10.1080/13554790903560422. Epub 2010 Feb 22. PMID 20178034
- [Background] Kuhn J, Lenartz D, Mai JK, Huff W, Lee SH, Koulousakis A, Klosterkoetter J, Sturm V. Deep brain stimulation of the nucleus accumbens and the internal capsule in therapeutically refractory Tourette-syndrome. J Neurol. 2007 Jul;254(7):963-5. doi: 10.1007/s00415-006-0404-8. Epub 2007 Apr 6. No abstract available. PMID 17410328
- [Background] Neuner I, Podoll K, Lenartz D, Sturm V, Schneider F. Deep brain stimulation in the nucleus accumbens for intractable Tourette's syndrome: follow-up report of 36 months. Biol Psychiatry. 2009 Feb 15;65(4):e5-6. doi: 10.1016/j.biopsych.2008.09.030. Epub 2008 Nov 12. No abstract available. PMID 19006786
- [Background] Zabek M, Sobstyl M, Koziara H, Dzierzecki S. Deep brain stimulation of the right nucleus accumbens in a patient with Tourette syndrome. Case report. Neurol Neurochir Pol. 2008 Nov-Dec;42(6):554-9. PMID 19235110
- [Background] Ackermans L, Temel Y, Cath D, van der Linden C, Bruggeman R, Kleijer M, Nederveen P, Schruers K, Colle H, Tijssen MA, Visser-Vandewalle V; Dutch Flemish Tourette Surgery Study Group. Deep brain stimulation in Tourette's syndrome: two targets? Mov Disord. 2006 May;21(5):709-13. doi: 10.1002/mds.20816. PMID 16463374
- [Background] Dehning S, Mehrkens JH, Muller N, Botzel K. Therapy-refractory Tourette syndrome: beneficial outcome with globus pallidus internus deep brain stimulation. Mov Disord. 2008 Jul 15;23(9):1300-2. doi: 10.1002/mds.21930. PMID 18528896
- [Background] Diederich NJ, Kalteis K, Stamenkovic M, Pieri V, Alesch F. Efficient internal pallidal stimulation in Gilles de la Tourette syndrome: a case report. Mov Disord. 2005 Nov;20(11):1496-9. doi: 10.1002/mds.20551. PMID 16037913
- [Background] Gallagher CL, Garell PC, Montgomery EB Jr. Hemi tics and deep brain stimulation. Neurology. 2006 Feb 14;66(3):E12. doi: 10.1212/01.wnl.0000190258.92496.a4. No abstract available. PMID 16476922
- [Background] Shahed J, Poysky J, Kenney C, Simpson R, Jankovic J. GPi deep brain stimulation for Tourette syndrome improves tics and psychiatric comorbidities. Neurology. 2007 Jan 9;68(2):159-60. doi: 10.1212/01.wnl.0000250354.81556.90. No abstract available. PMID 17210901
- [Background] Welter ML, Mallet L, Houeto JL, Karachi C, Czernecki V, Cornu P, Navarro S, Pidoux B, Dormont D, Bardinet E, Yelnik J, Damier P, Agid Y. Internal pallidal and thalamic stimulation in patients with Tourette syndrome. Arch Neurol. 2008 Jul;65(7):952-7. doi: 10.1001/archneur.65.7.952. PMID 18625864
- [Background] Martinez-Torres I, Hariz MI, Zrinzo L, Foltynie T, Limousin P. Improvement of tics after subthalamic nucleus deep brain stimulation. Neurology. 2009 May 19;72(20):1787-9. doi: 10.1212/WNL.0b013e3181a60a0c. No abstract available. PMID 19451536
- [Background] Karachi C, Grabli D, Baup N, Mounayar S, Tande D, Francois C, Hirsch EC. Dysfunction of the subthalamic nucleus induces behavioral and movement disorders in monkeys. Mov Disord. 2009 Jun 15;24(8):1183-92. doi: 10.1002/mds.22547. PMID 19412950
- [Background] Baup N, Grabli D, Karachi C, Mounayar S, Francois C, Yelnik J, Feger J, Tremblay L. High-frequency stimulation of the anterior subthalamic nucleus reduces stereotyped behaviors in primates. J Neurosci. 2008 Aug 27;28(35):8785-8. doi: 10.1523/JNEUROSCI.2384-08.2008. PMID 18753380
- [Background] Francois C, Grabli D, McCairn K, Jan C, Karachi C, Hirsch EC, Feger J, Tremblay L. Behavioural disorders induced by external globus pallidus dysfunction in primates II. Anatomical study. Brain. 2004 Sep;127(Pt 9):2055-70. doi: 10.1093/brain/awh239. Epub 2004 Aug 3. PMID 15292054
- [Background] Mallet L, Schupbach M, N'Diaye K, Remy P, Bardinet E, Czernecki V, Welter ML, Pelissolo A, Ruberg M, Agid Y, Yelnik J. Stimulation of subterritories of the subthalamic nucleus reveals its role in the integration of the emotional and motor aspects of behavior. Proc Natl Acad Sci U S A. 2007 Jun 19;104(25):10661-6. doi: 10.1073/pnas.0610849104. Epub 2007 Jun 7. PMID 17556546
- [Background] Ardouin C, Voon V, Worbe Y, Abouazar N, Czernecki V, Hosseini H, Pelissolo A, Moro E, Lhommee E, Lang AE, Agid Y, Benabid AL, Pollak P, Mallet L, Krack P. Pathological gambling in Parkinson's disease improves on chronic subthalamic nucleus stimulation. Mov Disord. 2006 Nov;21(11):1941-6. doi: 10.1002/mds.21098. PMID 16972268
- [Background] Houeto JL, Mallet L, Mesnage V, Tezenas du Montcel S, Behar C, Gargiulo M, Torny F, Pelissolo A, Welter ML, Agid Y. Subthalamic stimulation in Parkinson disease: behavior and social adaptation. Arch Neurol. 2006 Aug;63(8):1090-5. doi: 10.1001/archneur.63.8.1090. PMID 16908734
- [Background] Mallet L, Polosan M, Jaafari N, Baup N, Welter ML, Fontaine D, du Montcel ST, Yelnik J, Chereau I, Arbus C, Raoul S, Aouizerate B, Damier P, Chabardes S, Czernecki V, Ardouin C, Krebs MO, Bardinet E, Chaynes P, Burbaud P, Cornu P, Derost P, Bougerol T, Bataille B, Mattei V, Dormont D, Devaux B, Verin M, Houeto JL, Pollak P, Benabid AL, Agid Y, Krack P, Millet B, Pelissolo A; STOC Study Group. Subthalamic nucleus stimulation in severe obsessive-compulsive disorder. N Engl J Med. 2008 Nov 13;359(20):2121-34. doi: 10.1056/NEJMoa0708514. PMID 19005196
- [Background] Bohlhalter S, Goldfine A, Matteson S, Garraux G, Hanakawa T, Kansaku K, Wurzman R, Hallett M. Neural correlates of tic generation in Tourette syndrome: an event-related functional MRI study. Brain. 2006 Aug;129(Pt 8):2029-37. doi: 10.1093/brain/awl050. Epub 2006 Mar 6. PMID 16520330